CLINICAL TRIAL: NCT06053723
Title: The Effect of Bruxism on Masticatory Functionality and Severity of Temporomandibular Dsyfunction: A Cross-sectional Study
Brief Title: Bruxism and Severity of Temporomandibular Dsyfunction
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, Assist. Prof. Dr, Bandırma Onyedi Eylül University
Other Study IDs: 2023-54
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Temporomandibular Dysfunction
Keywords: temporomandibular dysfunction; bruxism; chewing functionality
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bruxism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fonseca's Anamnestic Questionnaire — The questionnaire includes 10 questions about joint, head and neck pain, pain during masticatory activity, parafunctional habits, decreased joint motion, impaired occlusion and emotional stress.
Other: Numeric Pain Scale — It is a simple, reliable and short-term method that is frequently used to measure pain intensity in the clinic.
Other: Jaw Functionality Limitation Scale-20 — It includes a total of 20 items, with "0" indicating no limitation and "10" indicating severe limitation in each item, about the function of the TMJ during different activities, difficulty in chewing and jaw limitation.

SUMMARY:
The aim of the study was to investigate the effect of bruxism on Temporomanbular joint functionality and dysfunction severity in individuals with Temporomandibular Dysfunction (TMD).

DETAILED DESCRIPTION:
The study included 91 individuals aged 20-55 years with TMD. Participants who volunteered to participate in the study signed the Informed Consent Form and completed the Descriptive Data Form including demographic characteristics. The presence of bruxism in individuals with TMD was questioned and the maximum mouth opening measurement was recorded. TMD severity was assessed by Fonseca's Anamnestic Questionnaire (FAQ), pain severity was assessed by Numeric Pain Scale (NPS), and masticatory and TMJ functioning was assessed by JAW Functional Limitation Scale-20 (JFLS-20). The evaluations of the participants were performed only once.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 55 years,
* Diagnosed with TMD,
* volunteer to participate in the study

Exclusion Criteria:

* having a non-reduced disc problem,
* surgical operation due to spine, abdomen and/or TMJ problem,
* trauma, cancer, neurological problems, congenital anomalies, musculoskeletal system problems,
* systemic disease,
* facial paralysis
* Less than 6 months of receiving any treatment related to the spine and TMJ

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: diagnosed with TMD
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Bruxism evaluation | April 2023- September 2023
  Sleep bruxism reported by the individual was recorded. As clinical diagnostic criteria for bruxism; the presence of regular or frequent teeth clenching and grinding sounds followed by pain or fatigue in the jaw muscles on waking up in the morning, temporal headache, masseter muscle hypertrophy, abnormal tooth abrasion and/or jaw locking were questioned and the presence of one or more clinical findings was recorded as bruxism.
Maximum mouth opening | April 2023- September 2023
  Maximum pain-free mouth opening was measured with a 15 cm ruler
Severity of Temporomandibular dysfunction | April 2023- September 2023
  Fonseca's Anamnestic Questionnaire (FAQ) was used. The questionnaire includes 10 questions about joint, head and neck pain, pain during masticatory activity, parafunctional habits, decreased joint motion, impaired occlusion and emotional stress. As a result of the questionnaire, the presence of TMD is accepted in patients with a score of 25 and above, and the severity can be classified as mild TMJ disorder (25-45), moderate TMJ disorder (50-65) and severe TMJ disorder (70-100).
Pain intensity | April 2023- September 2023
  Numeric Pain Scale (NAS): It is a simple, reliable and short-term method commonly used in the clinic to measure pain intensity. The patient is told that the most severe pain he/she feels in the TMJ region is 10, and if there is no pain, the pain intensity is 0. The participant was asked to say a number between 0 and 10 corresponding to the intensity of pain felt in the TMJ region.
Jaw Functionality | April 2023- September 2023
  Jaw Functionality Limitation Scale-20 was used. It includes a total of 20 items, with "0" indicating no limitation and "10" indicating severe limitation in each item, about the function of the TMJ during different activities, difficulty in chewing and jaw limitation. As a result of the questionnaire, it was reported that TMJ function was limited in individuals with a score of 5 and above.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Onyedi Eylul University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided